CLINICAL TRIAL: NCT05729906
Title: Dynamic Predictions of the Links Between Psychological and Physical Health of Older Patients in Nursing Home Via the Integration of "Multi-omics" Data.
Brief Title: Dynamic Predictions of the Links Between Psychological and Physical Health of Older Patients in Nursing Home
Acronym: BioMIND
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Research Center for Respiratory Diseases, Inserm U1100 (Unknown)
Responsible Party: Sponsor
Other Study IDs: DR220209-BioMIND
Record Dates: First submitted 2023-01-20; First posted 2023-02-15 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Psychological Health; Physical Health
Keywords: mental health; physical health; psychosomatic model; disability model; inflammation; metabolomics; nursing home; frailty; inflamm'aging
MeSH Terms: conditions — Psychological Well-Being; Inflammation; Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: psychological and physical tests — Once included (T0), participants will be reviewed at 6 (T1), and 12 (T2) months. At the three measurement times, research professionals (belonging to the PAVeA laboratory) will carry out, within the nursing home the physical and psychological measurements (classic standardized tests for the population). These measurements will be carried out in parallel with the routine biological explorations performed in the institution.
  At each visit, the remaining blood sampled in routine will be frozen in 2 aliquots for metabolomic and spectrometric analyses at the end of the study by the iBrain and Research Center for Respiratory Diseases laboratories.

SUMMARY:
Taking the older person as a whole is now essential to age well and prevent loss of functional independence. However, the relationship between physical and mental health remains not well understood. Combining the exploration of markers of inflammation, endocrine, nutritional, and metabolic functions, along with long-term monitoring of older persons, could allow for a comprehensive understanding of the biological phenotype, regardless of underlying pathologies. The primary objective will be to simultaneously test the psychosomatic model and the disability model in order to more fully account for the dynamic causal relationships between physical and mental health in older people. The investigators will investigate the mediating role of the biological phenotype on these relationships between mental and physical health. The independent and then combined analysis of specific candidate biomarkers will open up the possibility of identifying a biological mediation between mental and physical health. Furthermore, this will also allow us to deepen our understanding of the evolution of the immune-endocrine-metabolic state and, more broadly, of the biological phenotype of older people during aging.

DETAILED DESCRIPTION:
Promoting the health of older people to better support them remains one of the major challenges of the 21st century. More and more experts in gerontology (doctors, psychologists, sociologists, ...) are now advocating a holistic approach to older people. The recent recommendations of the WHO (2016) also invite us to favor an approach to aging centered on the potentialities and resources of older people more than on their deficiencies and diseases. Thus, taking into account the older person in his or her entirety ("body and mind") is a must for aging well and preventing the loss of functional independence. However, the relationship between physical and mental health remains poorly understood.

The psychosomatic model postulates that well-being and positive affects have an impact on physical health. It has thus been shown that good psychological health (e.g., positive mood, hope, optimism) has long-term beneficial effects on longevity, cardiovascular health, and chronic diseases. Conversely, poor mental health (e.g., presence of depressive symptoms) affects the health of older subjects and increases mortality risk. These results are in line with the so-called top-down approaches which postulate that well-being is a psychological trait that is the cause of future personal evaluations. In this psychosomatic approach, well-being, positive affect (i.e., good psychological health), is seen as antecedent to physical health. Naturally, it would seem unlikely that well-being would predict improved health for older people. However, well-being or the presence of positive affect could well predict different trajectories of "health" in ill older people.

In contrast, the so-called disability model postulates that physical health problems have an impact on psychological health, including well-being. This bottom-up approach considers physical health problems as antecedents of well-being. A study conducted by members of the laboratory supporting this project argues for this approach. The results show that poor physical health would unidirectionally predict poor life satisfaction over the long term.However, no study to date has been able to confirm the prevalence of one model over the other.

The main hypothesis of this research is based on the presence of a bi-directional pattern between physical and psychological health, and thus on the absence of a unique prevalence of one pattern over the other for the entire target elderly population. The investigators also hypothesize that the causal links between physical and psychological health may vary over time as a function of specific mediators, including inflammatory and metabolomic profiles. Our second hypothesis thus postulates that biological profiles could mediate the bi-directional links between physical and psychological health. For example, the investigators know that negative psychological affects have a negative impact on our "physical" health, so the investigators can assume that positive psychological affects can produce an anti-inflammatory effect, thus allowing us to be in better physical health (protective factor).

ELIGIBILITY:
Inclusion Criteria:

Institutionalized older adults over 65

Exclusion Criteria:

* older adults in palliative care
* older adults with severe cognitive impairment (MMSE <11)
* Opposition to data processing from the older adult or his/her guardian/trustee if under legal protection

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older persons over 65 in nursing homes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
PANAS | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Positive and Negative Affect Schedule (PANAS) (Caci & Bayle, 2007) to evaluate positive and negative affects (20 items with a 5-point Likert scale; a score /50 for negative affects, a score/50 for positive affects). In order to adapt to the possible cognitive disorders of the participants, they will be asked to answer on a visual analogical scale using the same rating as the initial scale (scale from 1 to 5, from "very little or not at all" to "very much").
PHQ-9 | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Patient Health Questionnaire (PHQ-9) (Kroenke et al., 2001) for thymia (9 items, 4-point Likert scale with a maximum score of 27). In order to adapt to the participants' possible cognitive disorders, they will be asked to answer on a visual analog scale using the same rating as the initial scale (scale from 0 to 3, from "never" to "almost every day").
Subjective Age Rating Scale | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  Subjective Age Rating Scale (1 item) to evaluate perceived age.
EVIBE (psychological) | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Instant Well-Being Rating Scale (EVIBE) (Delphin-Combe et al., 2018) is a scale to evaluate subjective psychological well-being (1-5 visual analog scale, a higher score means a better outcome).
MMSE | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Mini-Mental State Examination (MMSE) (Folstein et al. 1975) for global cognitive status (score from 0 to 30 points, a higher score means a better outcome). In order to most closely match the participant's cognitive abilities at each data collection time, MMSE scores will only be collected from the medical records if they are less than 2 months old.
SPPB | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Short Physical Performance Battery test (SPPB) (Guralnik et al., 2000) for overall physical ability (3 sub-scores on 4 points each [walking, strength, balance], score from 0 to 12, a higher score means a better outcome)
EVIBE (physical) | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Instant Well-Being Rating Scale (EVIBE) (Delphin-Combe et al., 2018) for subjective physical well-being (visual analog scale from 1 to 5, a higher score means a better outcome)
Diagnosis of undernutrition | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The questionnaire for the diagnosis of undernutrition according to HAS criteria, allowing the presence and degree of undernutrition to be assessed (13 items, the diagnosis of undernutrition requires the presence of at least: 1 phenotypic criterion and 1 etiological criteria. Undernutrition is qualified as severe if one of the criteria of severe undernutrition is verified) (HAS, 2021)
MNA | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Mini Nutritional Assessment (MNA) (Guigoz et al., 2006) for the nutritional profile (6 screening items - score frome 0 to 14 points, a higher score means a worse outcome)
Charlson score | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Charlson score (Charlson et al., 1987) for the collection of comorbidities (calculation of an index weighted according to age, a higher score means a worse outcome)
CIRS | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Cumulative Illness Rating Scale (CIRS) (Parmelee et al., 1995) for the collection of comorbidities (14 items evaluated from "none" to "very severe", score from 0 to 56, a higher score means a worse outcome).
ADLS | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  Activities of Daily Living Scale (ADLS) (Katz & Akpom, 1976) for the level of functional autonomy (6 items, score from 0 to 6, a higher score means a better outcome).
CFS | Evolution over time of the psychological health (T1-T0, T2-T1, T2-T0). T0: inclusion visit, T1: month 6 and T2: month 12.
  The Clinical Frailty Scale (CFS) (Abraham et al., 2019) for the evaluation of clinical frailty (only one item can be chosen, score from 1 to 9, a higher score means a worse outcome).

SECONDARY OUTCOMES:
inflammatory measures | T0: inclusion visit, T1: month 6 and T2: month 12
  * High Sensivity C-Reactive Protein (hsCRP)
  * Interleukins (IL-6, other IL) and pro- and anti-inflammatory mediators
  * Tumor Necrosis Factor-alpha (TNF-alpha)
  * Orosomucoid
  * Pre-albumin (Prognostic Inflammatory and Nutritional Index)
metabolomic profiles | T0: inclusion visit, T1: month 6 and T2: month 12
  Calculation of metabolite concentrations with metabolomic profile analyzed by high resolution mass spectrometry (LC/MS-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Wassim GANA, Principal Investigator — CHRU de Tours
Locations (5):
- France (5):
  - EHPAD CHIC Amboise/Chateau-Renault, Château-Renault
  - EHPAD Les Groussins, Chinon
  - EHPAD Paul Martinais, Loches
  - EHPAD Le Clos Mignot, Luynes
  - EHPAD l'Ermitage, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abraham P, Courvoisier DS, Annweiler C, Lenoir C, Millien T, Dalmaz F, Flaatten H, Moreno R, Christensen S, de Lange DW, Guidet B, Bendjelid K, Walder B, Bollen Pinto B. Validation of the clinical frailty score (CFS) in French language. BMC Geriatr. 2019 Nov 21;19(1):322. doi: 10.1186/s12877-019-1315-8. PMID 31752699
- [Background] Blazer DG, Hybels CF, Pieper CF. The association of depression and mortality in elderly persons: a case for multiple, independent pathways. J Gerontol A Biol Sci Med Sci. 2001 Aug;56(8):M505-9. doi: 10.1093/gerona/56.8.m505. PMID 11487603
- [Background] Boehm JK, Kubzansky LD. The heart's content: the association between positive psychological well-being and cardiovascular health. Psychol Bull. 2012 Jul;138(4):655-91. doi: 10.1037/a0027448. Epub 2012 Apr 16. PMID 22506752
- [Background] Brief AP, Butcher AH, George JM, Link KE. Integrating bottom-up and top-down theories of subjective well-being: the case of health. J Pers Soc Psychol. 1993 Apr;64(4):646-53. doi: 10.1037//0022-3514.64.4.646. PMID 8473981
- [Background] Caci, H., & Baylé, F. (2007). L'échelle d'affectivité positive et d'affectivité négative. Première traduction en français. Présenté au Congrès de l'Encéphale, Paris, 22-25.
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Chida Y, Steptoe A. Positive psychological well-being and mortality: a quantitative review of prospective observational studies. Psychosom Med. 2008 Sep;70(7):741-56. doi: 10.1097/PSY.0b013e31818105ba. Epub 2008 Aug 25. PMID 18725425
- [Background] Delphin-Combe F, Dauphinot V, Denormandie P, Sanchez S, Hay PE, Moutet C, Krolak-Salmon P. The Scale of instantaneous wellbeing: validity in a population with major neurocognitive disorders. Geriatr Psychol Neuropsychiatr Vieil. 2018 Sep 1;16(3):329-334. doi: 10.1684/pnv.2018.0745. PMID 30168440
- [Background] Gan Y. Happy People Live Longer and Better: Advances in Research on Subjective Well-Being. Appl Psychol Health Well Being. 2020 Mar;12(1):3-6. doi: 10.1111/aphw.12192. Epub 2020 Jan 29. No abstract available. PMID 31994837
- [Background] Diener E. Subjective well-being. Psychol Bull. 1984 May;95(3):542-75. No abstract available. PMID 6399758
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gana K, Bailly N, Saada Y, Joulain M, Trouillet R, Herve C, Alaphilippe D. Relationship between life satisfaction and physical health in older adults: a longitudinal test of cross-lagged and simultaneous effects. Health Psychol. 2013 Aug;32(8):896-904. doi: 10.1037/a0031656. Epub 2013 Mar 11. PMID 23477581
- [Background] Guigoz Y. The Mini Nutritional Assessment (MNA) review of the literature--What does it tell us? J Nutr Health Aging. 2006 Nov-Dec;10(6):466-85; discussion 485-7. PMID 17183419
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Hernandez R, Bassett SM, Boughton SW, Schuette SA, Shiu EW, Moskowitz JT. Psychological Well-being and Physical Health: Associations, Mechanisms, and Future Directions. Emot Rev. 2018 Jan;10(1):18-29. doi: 10.1177/1754073917697824. Epub 2017 Oct 20. PMID 36650890
- [Background] Katz S, Akpom CA. A measure of primary sociobiological functions. Int J Health Serv. 1976;6(3):493-508. doi: 10.2190/UURL-2RYU-WRYD-EY3K. PMID 133997
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Parmelee PA, Thuras PD, Katz IR, Lawton MP. Validation of the Cumulative Illness Rating Scale in a geriatric residential population. J Am Geriatr Soc. 1995 Feb;43(2):130-7. doi: 10.1111/j.1532-5415.1995.tb06377.x. PMID 7836636